CLINICAL TRIAL: NCT01447329
Title: Ear Acupuncture for Post-operative Pain Associated With Ambulatory Arthroscopic Knee Surgery - A Randomized Controlled Trial
Brief Title: Ear Acupuncture for Pain Associated With Ambulatory Arthroscopic Knee Surgery
Acronym: BFAKnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20110169H
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pain
Keywords: pain; acupuncture; knee; debridement; surgery; arthroscopic knee surgery debridement
MeSH Terms: conditions — Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment plus ear acupuncture (Experimental): Standard treatment plus ear acupuncture
  Interventions: Other: Ear Acupuncture
- standard (Placebo Comparator): placebo
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Other: Ear Acupuncture — Ear acupuncture utilizes up to 10 needles. The ear Acupuncture points on the right ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero. The ear Acupuncture points on the left ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero. The subject will receive five needles intra-operatively on each ear.
  Other Names: Sedatelec ASP Original Gold needles
  Arms: Standard treatment plus ear acupuncture
Drug: Standard Treatment
  Arms: standard

SUMMARY:
The investigators propose to complete a randomized controlled trial to compare ear acupuncture at Cingulate gyrus, thalamus, omega 2, shen-men, and point zero on the right and left ear plus standard of care versus standard of care alone for symptomatic treatment of pain following ambulatory arthroscopic knee surgery. After the subject has been discharged, phone calls, emails or text messages will be made at 24 and 48 hours, 1 week and 1 month. These contacts will be used to assess the subject's pain level, ambulation status, doses of analgesics taken and time to return to full duty. At 1 week and 1 month, subjects will be asked the PIQ-6 Pain Impact Questionnaire.

DETAILED DESCRIPTION:
Subjects (DoD beneficiaries) that are 18 years or older with a scheduled ambulatory arthroscopic knee surgery will present for their pre-op appointment. At the time of check-in the subjects meeting the inclusion criteria, will be offered the opportunity to participate. Informed Consent and HIPAA Authorization will be obtained prior to any study-related procedures or any sedation being performed. The subject will be asked the screening questions for exclusion criteria (See attached instrument). The PI will have the AI or Study staffs recruit their patients to prevent any misconception of coercion. The subjects Armed Forces Health Longitudinal Technology Application (AHLTA) record including previous encounters, vital signs review, medication list, demographics and problems list will be reviewed by one of the investigators to confirm the inclusion/exclusion criteria have been met. The investigator will evaluate the subject and determine any further exclusion criteria based on exam. These subjects will then be randomized into two groups using a random number generator via block randomization by the Research Coordinator:

Group 1: Standard treatment alone Group 2: Standard treatment plus ear acupuncture

Subjects will be asked upon admittance to the PACU and the SDSU to answer the questions in the Data Collection Tool. Subjects will be given treatment while in the operating room and while under sedation according to their randomization group. The right and left ears will be cleansed with an alcohol swab prior to ear acupuncture. All subjects, regardless of study group, will get band aid to cover both ears. This is done to blind the orthopedic surgeon, the anesthesiologist and any nursing staff that comes in contact with the patient. Even though they are getting standard of care pain treatment, the investigators are blinding these individuals to remove any potential of bias when they are assessing a subject's pain. Subjects in both groups will be instructed to remove the band aids 24 hours after their surgery. After the subject has been discharged, phone calls, emails or text messages will be made at 24 and 48 hours, 1 week and 1 month. These contacts will be used to assess the subject's pain level, ambulation status, doses of analgesics taken and time to return to full duty. At 1 week and 1 month, subjects will be asked the PIQ-6 Pain Impact Questionnaire.

Subjects are getting the knee arthroscopy as part of standard of care in this study. It is standard of care to have military members return to to light-duty 2 weeks after knee arthroscopy and full-duty 6 weeks after knee arthroscopy. Should the subject return to duty with the acupuncture needles still in place, this will not affect their ability to perform their duties, however, to maintain compliance with AFI 36-2903, you may want to remove the needles or place a bandage over both ears to cover the ear acupuncture needles.

Ear acupuncture utilizes up to 10 needles. The ear Acupuncture points on the right ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero. The ear Acupuncture points on the left ear include Cingulate gyrus, thalamus, omega 2, shen-men, point zero. The subject will receive five needles intra-operatively on each ear.

Subject's participation in this study is completed after 1 month.

Patients in group 2 who are receiving ear Acupuncture will be instructed to have no heavy meals, excessive hot or cold foods, heavy exercise or intercourse and no alcohol for 24 hours. Ear Acupuncture needles will fall out on their own within about 6 days.

All investigators are trained in Battlefield Acupuncture and credentialed by the MOFH Credentials committee to perform Battlefield Acupuncture.

The investigators anticipate that the ear acupuncture will reduce the doses of analgesics needed to control pain, decrease time to discharge, reduce time to ambulation without assistance and improve return to duty time.

The standing orders for post-operative care pain control are attached. The risks associated with the use of ear acupuncture needles include: pain, bleeding, infection (very rare) and flare of signs and symptoms. In the event the acupuncture needles do not fall out within 6 days, patients will be instructed to come in and have them removed by one of the Investigators. In this study the investigators are using Sedatelec ASP Original Gold needles. These acupuncture needles are sterile, gold plated semi permanent ear acupuncture needles for single use.

If at any time during the study, the subject decides to withdraw from the study, they can come in and have the ear acupuncture needles removed by one of the Investigators. If patients are withdrawn from the study, they will have the option to either have the acupuncture needles removed by one of the investigators or allow them to fall out on their own.

Patients must agree to take precautions to prevent pregnancy during the initial phase (surgery) of this study. Pregnancy tests are routinely done as standard of care for all women prior to surgery. The only completely reliable methods of birth control are total abstinence or surgical removal of the uterus. Other methods, such as the use of condoms, a diaphragm or cervical cap, birth control pills, IUD, or sperm killing products are not totally effective in preventing pregnancy. Also, women who are breastfeeding at the time of surgery may not participate in this study.

ELIGIBILITY:
Inclusion:

* Tricare beneficiaries receiving care at Nellis AFB.
* Male and female subjects (DoD beneficiaries), 18 years or older scheduled for ambulatory unilateral arthroscopic knee surgery.
* Unilateral arthroscopic knee surgery debridement.

Exclusion:

* History of significant gastrointestinal bleed
* Previous documented history of stage 2 kidney disease or worse
* Pregnant or breastfeeding
* History of gastric bypass surgery
* Chronic oral steroids use
* Absence of ear
* Active cellulitis of ear
* Ear anatomy precluding identification of acupuncture landmarks
* Non-English speaking
* Taking Coumadin or any Heparin-based anticoagulant
* Use of Hearing Aids that preclude the insertion of ASP needles
* Allergy to study medications
* Inability to comply with study protocol
* Arthroscopic knee surgery with ligamentous repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Moss, M.D. Capt, Principal Investigator — Mike O'Callaghan Federal Hospital/Nellis AFB
Locations (1):
- Mike O'Callaghan Federal Hospital, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard: placebo
  Standard Treatment
Period: Overall Study
Arm/Group | Standard Treatment Plus Ear Acupuncture | Standard
Started | 24 | 25
Completed | 18 | 16
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Plus Ear Acupuncture | Standard | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants] — Population: Overall recruited versus overall analyzed.
  Participants
    number analyzed (Participants) | 18 | 16 | 34
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 18 | 16 | 34
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in Pain Level
Time Frame: during PACU (Post Anesthesia Care Unit) and SDSU (Same Day Surgical Unit) admissions, 24 and 48 hours, 1 week and 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Plus Ear Acupuncture | Standard
Number analyzed (Participants) | 24 | 25
Participants | 18 | 16

2. Primary Outcome: Ability to Ambulate Without Assistance
Time Frame: during PACU (Post Anesthesia Care Unit) and SDSU (Same Day Surgical Unit), 24 and 48 hours, 1 week and 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Plus Ear Acupuncture | Standard
Number analyzed (Participants) | 24 | 25
Participants | 18 | 16

3. Primary Outcome: Number of Patients With Reduced Analgesic Use
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Plus Ear Acupuncture | Standard
Number analyzed (Participants) | 24 | 25
Participants | 18 | 16

ADVERSE EVENTS:
Arm/Group | Standard Treatment Plus Ear Acupuncture | Standard
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes